CLINICAL TRIAL: NCT02732392
Title: Validation of Radioisotope Guided Lymphadenectomy for Loco-regional Staging in Patients With Intermediate or High-risk Prostate Cancer
Acronym: SENTINELLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2012-07; 2012-A-000287-36 (Registry Identifier: ID RCB)
Record Dates: First submitted 2016-03-30; First posted 2016-04-08 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: Patient With Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lymphadenectomy (Experimental)
  Interventions: Procedure: standard lymphadenectomy; Procedure: lymphadenectomy radio-isotope method

INTERVENTIONS:
Procedure: standard lymphadenectomy
Procedure: lymphadenectomy radio-isotope method

SUMMARY:
The diagnosis of a ganglionic infringement(achievement) at a patient reached (affected) by a prostate cancer is a factor(mailman) of bad forecast. The locoregional ganglionic staging is a very important element in the coverage (care). He allows to determine the local extension of the disease and the type(chap) of therapeutics to implement(operate) after the surgery. The standard cleaning out at present recommended by the European company (society) of urology at the patients at intermediate or high risk of second offense (recurrence) after local treatment(processing), has to concern the obturating pit, the internal and external iliac territories. However this type(chap) of cleaning out does not seem to solve all the problems of locoregional stratification. Indeed, several studies concerning the radio-controlled cleaning out highlighted that 10 in 30% of ganglions.

ELIGIBILITY:
Inclusion Criteria:

* Subject man, whose age is greater than or equal to 18 years
* Carrier of cancer intermediate risk non-metastatic prostate or high relapse
* Subject with an initial balance sheet expansion, regional and general negative by Scanner, abdominopelvic MRI or bone scan,
* Subject has undergone a medical examination in connection with the study,
* Topic for which a radical prostatectomy is considered curative purposes,
* Supported by Subject surgical teams involved in the study,
* Topic affiliated to a social security scheme,
* Subject who signed informed consent.

Exclusion Criteria:

* Subject man, whose age is less than 18 years
* Subject who have received hormone therapy or radiation therapy for prostate cancer
* Subject who had surgery for prostate adenoma (transurethral resection or open surgery) because of potential difficulties injection of radioactive tracer in the gland,
* Subject has a history of pelvic surgery or radiotherapy,
* Subject with inguinal hernia repair history of laparoscopic,
* Subject refusing blood transfusions,
* Subject is not agreeing to participate in this study and did not sign the informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2013-01-09 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2023-04-07 (Actual)

PRIMARY OUTCOMES:
Number of sentinel nodes radiolabeled | 54 months
  Number of sentinel nodes radiolabeled radiolabeled in the area of standard cleaning
Number of sentinel nodes radiolabeled | 54 months
  Number of sentinel nodes radiolabeled outside the standard cleaning of territory

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Lannes F, Baboudjian M, Ruffion A, Rouy M, Giammarile F, Rousseau T, Kraeber-Bodere F, Rousseau C, Rusu D, Colombie M, Brenot-Rossi I, Rossi D, Mottet N, Bastide C. Radioisotope-guided Lymphadenectomy for Pelvic Lymph Node Staging in Patients With Intermediate- and High-risk Prostate Cancer (The Prospective SENTINELLE Study). J Urol. 2023 Feb;209(2):364-373. doi: 10.1097/JU.0000000000003043. Epub 2022 Nov 4. PMID 36331157